CLINICAL TRIAL: NCT01415180
Title: Life After Pediatric Sepsis Evaluation
Acronym: LAPSE
Status: Completed | Type: Observational
Sponsor: Seattle Children's Hospital (Other)
Collaborators: The National Collaborative Pediatric Critical Care Research Network (Network); Children's Hospital Los Angeles (Other); Children's Hospital of Michigan (Other); Children's Hospital of Philadelphia (Other); University of Pittsburgh (Other); University of California, Los Angeles (Other); C.S. Mott Children's Hospital (Other); Children's National Research Institute (Other); Phoenix Children's Hospital (Other); Texas A&M University (Other)
Responsible Party: Principal Investigator, Jerry Zimmerman, Principal Investigator, Seattle Children's Hospital
Other Study IDs: SeattleChildrens
Record Dates: First submitted 2011-08-10; First posted 2011-08-11 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Septic Shock
Keywords: sepsis; health related quality of life; functional status; chronic comorbid conditions; organ dysfunction
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: previously healthy: Previously healthy children, without chronic disease prior to the sepsis episode, expected to comprise about 50-60% of the total study population.
- Children: chronic, complex conditions: Children with chronic, complex conditions prior to the sepsis episode, expected to comprise about 40-50% of the study population.

SUMMARY:
Sepsis represents the leading cause of childhood mortality worldwide. However, as distinct from adult medicine, there exists a large knowledge gap regarding long term health related quality of life (HRQL) and functional status (FS) following pediatric sepsis. This lack of sepsis outcomes data is critical because failure to identify children at risk for sepsis associated HRQL/FS deterioration may delay delivery of crucial rehabilitation medicine efforts to facilitate recovery. Moreover, failure to identify mechanisms of sepsis associated HRQL/FS deterioration may impede development of novel, effective interventions for these children. For the first time the LAPSE investigation will quantify deterioration of HRQL/FS among children surviving sepsis. We will measure the incidence, magnitude and duration of HRQL/FS alterations associated with pediatric septic shock, and examine clinical, sociodemographic, and parent/family factors potentially associated with such adverse outcomes. Because sepsis affects a heterogeneous group of children, long term morbidity associated with sepsis likely depends on premorbid health status and parent, family and home characteristics, as well as children's clinical course during sepsis critical illness. Mechanisms underlying adverse sepsis outcomes among children are poorly understood at this time. Clinically multiple organ dysfunction syndrome (MODS) has been clearly linked to sepsis mortality. To begin to understand pathophysiology underlying pediatric sepsis morbidity, this investigation will seek to identify evidence for association of HRQL/FS alterations following sepsis with intensity and duration of sepsis mediated organ dysfunction as well as with pre-existing comorbidities and parent, family, and home characteristics. The long-term goal of this research program is to timely identify children at high risk of sepsis mediated HRQL/FS deterioration and ultimately to design effective interventions to minimize such risk. The primary objectives of this investigation are to comprehensively characterize HRQL/FS trajectory and to critically examine the potential role of sepsis mediated organ dysfunction as well as pre-existing comorbidities and parent, family, and home characteristics as risk factors for the adverse outcomes. The central hypothesis is that intensity of sepsis organ dysfunction will predict magnitude of HRQL/FS deterioration. We also hypothesize that the trajectory towards baseline HRQL/FS following the sepsis event will also depend on pre-existing co-morbidities and parent, family, and home, and characteristics. Knowledge of these potential mechanisms will ultimately facilitate development of targeted interventions to maximize HRQL/FS among children surviving sepsis.

DETAILED DESCRIPTION:
In-hospital pediatric sepsis mortality has decreased substantially, but long-term mortality and morbidity among children initially surviving sepsis, is unknown. Accordingly, the Life After Pediatric Sepsis Evaluation investigation was conducted to describe the trajectory of mortality and health-related quality of life morbidity and critical illness factors associated with these outcomes for children encountering community-acquired septic shock.

Design: Prospective, cohort-outcome study, conducted 2013-2017. Setting: Twelve academic pediatric intensive care units (PICUs) in the United States.

Patients: Critically ill children, 1 month to 18 years, with community-acquired septic shock requiring vasoactive-inotropic support. Interventions: Demographic, infection, and illness severity data were collected at PICU admission. Organ dysfunction and resource utilization data were collected during PICU stay. Serial parent proxy-report health-related quality of life assessments were obtained at baseline, 7 days, and 1, 3, 6, and 12 months following PICU admission utilizing the Pediatric Quality of Life Inventory or Stein-Jessop Functional Status Scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 44 weeks EGA to 18 years
* Admitted to the PICU for the sepsis event
* Evidence of SIRS including fever/ hypothermia and leukocytosis/leukopenia
* Documented or suspected infection
* Cardiovascular organ dysfunction with need for vasoactive-inotropic support

Exclusion Criteria:

* Lack of commitment to aggressive sepsis therapy OR
* Ward of the state OR
* Sepsis event associated with a PICU-acquired nosocomial infection OR
* Parents do not speak English or Spanish OR
* Previously enrolled in the LAPSE study
* Enrollment not possible within 12 hours of PICU admission

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 0-18 admitted to a PICU for septic shock
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Specific Aim 1: Measure alterations in HRQL/FS longitudinally among children with septic shock. | Baseline, PICU discharge, 1, 3, 6, 12 months following PICU admission for sepsis
  Hypotheses related to this specific aim include:
  1.1 A majority of children with septic shock will demonstrate declination of generic HRQL/FS comparing baseline and one month post-enrollment measures. [Incidence]
  1.2 Significant deterioration in generic HRQL/FS will occur among children with septic shock comparing baseline and one month post-enrollment measures. [Magnitude]
  1.3 Normalization of HRQL/FS will be observed by 12 months for the majority of children surviving septic shock. [Duration]

SECONDARY OUTCOMES:
Specific Aim 2: Determine the association between the magnitude of septic shock related HRQL/FS deterioration with validated measures of sepsis-mediated organ dysfunction. | Baseline, PICU discharge, 1, 3, 6, 12 months following PICU admission for sepsis
  Hypotheses related to this specific aim include:
  2.1 Magnitude of septic shock related generic HRQL/FS deterioration will be associated with area under the curve of validated organ dysfunction measures assessed daily during PICU stay for the sepsis event.
Specific Aim 3: Describe the association between longitudinal changes in HRQL/FS following septic shock with measures of parent, family, and home characteristics and pre-existing comorbidities. | Baseline, PICU discharge, 1, 3, 6, 12 months following PICU admission for sepsis
  Hypotheses related to this specific aim include:
  3.1 Family and home characteristics (socio-economic status, parental educational attainment, family function, parental distress, and insurance status) will be associated with duration and magnitude of HRQL/FS alterations.
  3.2 Complexity of chronic comorbid conditions will be associated with duration and magnitude of HRQL/FS alterations

CONTACTS AND LOCATIONS:
Overall Officials: Jerry J. Zimmerman, MD, PhD, Principal Investigator — Seattle Children's Hospital
Locations (11):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Mattel Children's Hospital, Los Angeles, California
  - National Children's Hospital, Washington D.C., District of Columbia
  - Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pittsburgh Children's Hospital, Pittsburgh, Pennsylvania
  - Texas A&M University, College Station, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Result] Zimmerman JJ, Banks R, Berg RA, Zuppa A, Newth CJ, Wessel D, Pollack MM, Meert KL, Hall MW, Quasney M, Sapru A, Carcillo JA, McQuillen PS, Mourani PM, Wong H, Chima RS, Holubkov R, Coleman W, Sorenson S, Varni JW, McGalliard J, Haaland W, Whitlock K, Dean JM, Reeder RW; Life After Pediatric Sepsis Evaluation (LAPSE) Investigators. Critical Illness Factors Associated With Long-Term Mortality and Health-Related Quality of Life Morbidity Following Community-Acquired Pediatric Septic Shock. Crit Care Med. 2020 Mar;48(3):319-328. doi: 10.1097/CCM.0000000000004122. PMID 32058369
- [Result] Zimmerman JJ, Banks R, Berg RA, Zuppa A, Newth CJ, Wessel D, Pollack MM, Meert KL, Hall MW, Quasney M, Sapru A, Carcillo JA, McQuillen PS, Mourani PM, Wong H, Chima RS, Holubkov R, Coleman W, Sorenson S, Varni JW, McGalliard J, Haaland W, Whitlock K, Dean JM, Reeder RW; Life After Pediatric Sepsis Evaluation (LAPSE) Investigators. Trajectory of Mortality and Health-Related Quality of Life Morbidity Following Community-Acquired Pediatric Septic Shock. Crit Care Med. 2020 Mar;48(3):329-337. doi: 10.1097/CCM.0000000000004123. PMID 32058370
- [Result] Meert KL, Reeder R, Maddux AB, Banks R, Berg RA, Zuppa A, Newth CJ, Wessel D, Pollack MM, Hall MW, Quasney M, Sapru A, Carcillo JA, McQuillen PS, Mourani PM, Chima RS, Holubkov R, Sorenson S, Varni JW, McGalliard J, Haaland W, Whitlock KB, Dean JM, Zimmerman JJ; and the Life After Pediatric Sepsis Evaluation (LAPSE) Investigators. Trajectories and Risk Factors for Altered Physical and Psychosocial Health-Related Quality of Life After Pediatric Community-Acquired Septic Shock. Pediatr Crit Care Med. 2020 Oct;21(10):869-878. doi: 10.1097/PCC.0000000000002374. PMID 32667767
- [Result] Murphy LK, Palermo TM, Meert KL, Reeder R, Dean JM, Banks R, Berg RA, Carcillo JA, Chima R, McGalliard J, Haaland W, Holubkov R, Mourani PM, Pollack MM, Sapru A, Sorenson S, Varni JW, Zimmerman J. Longitudinal Trajectories of Caregiver Distress and Family Functioning After Community-Acquired Pediatric Septic Shock. Pediatr Crit Care Med. 2020 Sep;21(9):787-796. doi: 10.1097/PCC.0000000000002404. PMID 32541376
- [Result] Starr MC, Banks R, Reeder RW, Fitzgerald JC, Pollack MM, Meert KL, McQuillen PS, Mourani PM, Chima RS, Sorenson S, Varni JW, Hingorani S, Zimmerman JJ; Life After Pediatric Sepsis Evaluation (LAPSE) Investigators. Severe Acute Kidney Injury Is Associated With Increased Risk of Death and New Morbidity After Pediatric Septic Shock. Pediatr Crit Care Med. 2020 Sep;21(9):e686-e695. doi: 10.1097/PCC.0000000000002418. PMID 32569242